CLINICAL TRIAL: NCT00674765
Title: A Phase II Double-blind, Placebo-controlled Trial of Quetiapine for Frequent, Heavy Drinkers (Seroquel2)
Brief Title: Seroquel for Frequent, Heavy Drinkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 807057 - Kampan_AA016553; NIH Grant 1R01AA016553-01A1
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Seroquel
  Interventions: Drug: Seroquel
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seroquel — 400 mg/day
  Other Names: quetiapine
  Arms: 1
Drug: Placebo — 400 mg/day
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effects of quetiapine in reducing percent heavy drinking days and increasing percent abstinent days in alcohol dependent patients who are frequent heavy drinkers.

DETAILED DESCRIPTION:
This trial is a phase 2, randomized, double-blind, placebo-controlled, parallel group trial intended to assess the efficacy of quetiapine compared to placebo in alcoholics who are frequent heavy drinkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, 18-70 years old.
2. Meets DSM-IV criteria for current diagnoses of alcohol dependence, determined by the MINI/SCID-IV {First, 1996 #34}.
3. Meets the drinking criteria, measured by TLFB and the Addiction Severity Index {McLellan, 1992 #37}:
4. Three consecutive days of abstinence from alcohol immediately before randomization
5. Lives a commutable distance from the TRC and agrees to attend all research visits including follow-up visits.
6. Speaks, understands, and prints in English.

Exclusion Criteria:

1. Has evidence of dependence on a substance other than alcohol (except nicotine and marijuana).
2. Tests positive on the urine drug screen during the screening weeks (one retest allowed). Subjects whose urine drug screen tests positive for benzodiazepines will be allowed to randomize, at the discretion of the PI, if they are known to be physician-prescribed for detox purposes.
3. Has hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) of at least 4.5 times normal after the required 3 days of abstinence, or elevated bilirubin (>1.3), with associated elevations of AST and ALT above normal limits.
4. Meets diagnostic criteria for a current unstable or serious psychiatric or medical illness.

   Has serious heart, lung, kidney, immune system, GI tract (ulcerative colitis, regional enteritis, or gastrointestinal bleeding) disease.
5. Has taken any psychotropic medications (including disulfiram, naltrexone or acamprosate) regularly within the last 2 weeks or needs immediate treatment with a psychotropic medication.
6. Tests positive on a pregnancy test, is contemplating pregnancy in the next 12 months, is nursing, or is not using an effective contraceptive method if the patient is of child-bearing potential, meaning has not had a hysterectomy or is in menopause, meaning 50 or over and has not had a menstrual cycle in 12 months.
7. Has known hypersensitivity to antipsychotics.
8. Has taken any investigational drug as part of an investigational trial within 30 days prior to the randomization.
9. A history of seizure disorder.
10. The presence of cataracts.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Kampman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Seroquel: Seroquel
  Seroquel: 400 mg/day
- Placebo: Placebo
  Placebo: 400 mg/day
Period: Overall Study
Arm/Group | Seroquel | Placebo
Started | 81 | 75
Completed | 45 | 46
Not Completed | 36 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seroquel | Placebo | Total
Number analyzed (Participants) | 81 | 75 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (9.9) | 45.4 (11.3) | 44.4 (10.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 75 | 156
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 65 | 60 | 125
Region of Enrollment [Number; unit: participants]
  United States | 81 | 75 | 156

OUTCOME MEASURES:

1. Primary Outcome: TimeLine Follow Back (TLFB) to Measure Percent Heavy Drinking Days During the Medication/Placebo Phase
Description: The total number of heavy drinking days per Arm was divided by total number of days, multiplied by 100%, to report the percent days of heavy drinking per Arm.
Time Frame: 12 weeks
Measure: Number; unit: percent days of heavy drinking
Groups:
- Seroquel (Quetiapine): Seroquel (quetiapine)
  Seroquel: 400 mg/day
- Placebo Sugar Pill: Placebo
  Placebo: 400 mg/day
Arm/Group | Seroquel (Quetiapine) | Placebo Sugar Pill
Number analyzed (Participants) | 81 | 75
percent days of heavy drinking | 20 | 24
Statistical Analysis 1: Comparison: Seroquel (Quetiapine) vs Placebo Sugar Pill; Test type: Superiority or Other; p = .388, t-test, 2 sided; t=.87

ADVERSE EVENTS:
Arm/Group | Seroquel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/75
Other Adverse Events (participants affected / at risk) | 76/81 | 41/75
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Seroquel (N=81) | Placebo (N=75)
Sedation (General disorders) | 43 | 22
Dry Mouth (General disorders) | 16 | 6
Increased appetite (Metabolism and nutrition disorders) | 13 | 6
Headache (General disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes